CLINICAL TRIAL: NCT04371432
Title: Genetics of COVID-19 Susceptibility and Manifestations
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200090; 20-HG-0090
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: COVID-19; Coronavirus 2019
Keywords: SARS-CoV-2; Whole Exome Sequencing; Coronavirus 2019; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sample Group 1 (NIHCC): Existing NIH Clinical Center patients/participants tested positive for SARS-CoV-2 invited to participate by their NIH study team
- Sample Group 2 (OMS & Field): Recruited through NIH OMS, referred by collaborators or who self-refer, tested positive for SARS-CoV-2 (and selected relatives of participants irrespective of infection status)

SUMMARY:
Background:

Coronavirus 2019 (COVID-19, or SARS-CoV-2) is a serious public health problem, and genetics may play a role in how serious the illness becomes in certain people. Genes are the instructions that our body uses to grow and develop. Variations in our genes can cause medical conditions and may be the reason why some people get sicker than others.

Objective:

This study aims to learn more about the genetic contributions to the severity of COVID-19. We hope to use this information to develop therapies that reduce the severity of COVID-19 symptoms in some people.

Eligibility:

Anyone located in the United States who has tested positive for SARS-CoV-2 infection may be eligible to join (including NIH staff).

Design:

Participants will complete a questionnaire about their health history and COVID-19 symptoms.

Participants will give a blood or saliva sample. It will be about 2 tablespoons of blood, or we will send a saliva collection kit. Researchers will use this blood or saliva sample to study the participant s DNA.

The data about participants genes will be stored in a large database. The database will be shared with other qualified researchers who are trying to learn about COVID-19. Participants names and other personal details will not be shared. Instead, the data will be labeled with a code.

Participants may be contacted by study team members for up to a year after they join the study.

DETAILED DESCRIPTION:
The current SARS-CoV-2 pandemic presents a serious challenge to public health. Individuals infected with SARS-CoV-2 experience extremes in symptomatology ranging from a complete lack of symptoms to rapidly worsening end-stage pulmonary disease. The explanatory mechanism underlying susceptibility to severe disease remains unknown. We hypothesize that underlying genetic factors are at least partially explanatory. We aim to employ a phenotypic extremes approach to rapidly ascertain severely and mildly affected COVID-19 patients for genomic interrogation to identify germline and somatic variants that may play a role in host susceptibility to disease to correlate those phenotypic extremes with genetic variants. We will employ both a rare and common variant approach, using both genome sequencing and SNP chip analysis and B and T cell repertoire interrogation.

ELIGIBILITY:
* INCLUSION CRITERIA
* Cohort 1 (Existing NIH Clinical Center Patient/Participants invited to participate by their NIH study team)
* Cohort 2 (Individuals recruited through NIH Occupational Medicine Services (OMS) patients referred by NIH investigators or other providers; individuals who self-refer)
* Located in the United States
* Positive test for SARS-CoV-2 virus infection
* Age greater than or equal to 3 years old

  * only for participants providing a blood sample

EXCLUSION CRITERIA:

* Individuals for whom we cannot consent for participation in a language offered by our existing interpretation service.
* Weight less than 10 kg*

Ages: 1 Month to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This protocol will only enroll identifiable participants by invitation only. De-identified biospecimens and/or other clinical information may be analyzed. All prospective study participants will be notified of their potential eligibility by an established contact at the NIH Clinical Center. Cohort 1= Existing NIH Clinical Center inpatients/participants tested positive for SARS-CoV-2 invited to participate by their NIH study team; Cohort 2= Individuals recruited through NIH OMS, patients referred by collaborators, patients who self-refer, tested positive for SARS-CoV-2 with mild or severe manifestations of COVID-19 disease (and selected relatives of participants irrespective of infection status)
Sampling Method: Non-Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Molecular etiology of host susceptibility to severe COVID-19 | Ongoing
  Identify common and rare germline variants associated with host susceptibility to severe or fatal COVID-19 disease using a case-case design.

SECONDARY OUTCOMES:
Mechanisms of disease | Ongoing
  Perform exploratory analyses of epigenetic signatures, serologic immune markers and antibody profiles, and other possible techniques to discover other mechanisms of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie G Biesecker, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be deposited into the database of genotypes and phenotypes (dbGaP), which is designed with tiered access to clinical data. There is open, public access to summary clinical data of study participants and qualified investigators may apply for access to individual, coded clinical results. Access is limited to authorized medical researchers and redistribution and security policies are strict. Broad future use of data deposited into dbGaP will be permitted.@@@De-identified data will be made available to collaborators. As members of the COVID-19 Host Genetics Initiative and we will collaborate and share data on rare variant analyses with the consortium, per NIH policy.@@@This study will comply with the NIH GDS Policy.@@@Samples and/or data may be shared with other researchers in coded form if their studies relate to the broadly defined purpose of increasing the understanding of the genetic contributions to disease expression of COVID-19, per NIH policy.@@@
Supporting Information: Study Protocol
Time Frame: IPD will be shared per NIH policy and available through the closure of the study. At the time the study is closed, a proposal to the IRB will be made to keep the data or destroy it.
Access Criteria: dbGap is a controlled-access database with view-only access to summary-level information and individual-level genotype and sequence data associated with phenotypic features. @@@De-identified data from this study will be made available to collaborators and as members of the COVID-19 Host Genetics Initiative and we will extensively collaborate and share data on rare variant analyses with the consortium, per NIH policies on Genomic Data Sharing.@@@This study will comply with the NIH Genomic Data Sharing Policy, which applies to all NIH-funded research that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data.@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-HG-0090.html